CLINICAL TRIAL: NCT04408131
Title: Morbi-mortality by COVID-19 Among Homeless People in Marseille: a Cohort Study
Acronym: COVIDHomeless
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study not started
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-32; 2020-A01398-31 (Other: ID RCB)
Record Dates: First submitted 2020-05-28; First posted 2020-05-29 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Homeless
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Homeless people (Experimental): Blood sample
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — virological test
Biological: Blood sample — serological test

SUMMARY:
COVID/Homeless is a prospective observational cohort study of homeless people to determine the impact of the SARS-CoV-2 epidemic on this population.

The cohort aims for exhaustiveness for the city of Marseille, being based on the active files of the partner teams, namely the four emergency shelters of Marseille and 12 outreach teams (including one specialized in psychiatry, three specialized in addictions, and three working in squats and shantytowns).

Aims of this cohort include to identify of the prognostic factors of morbi-mortality of homeless people by COVID-19, and therefore to propose appropriate management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Living in the city of Marseille
* Being homeless
* Be over 18 years of age

Exclusion Criteria:

* Persons under guardianship
* Persons who refused to sign the research consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-01-27 (Estimated); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
the covid mortality rate | 90 days
  The mortality rate is determined by the initial clinical diagnosis and follow-up of the patient by the field team.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mosnier E, Loubiere S, Monfardini E, Alibert A, Landier J, Ninoves L, Bosetti T, Auquier P, Mosnier M, Wakap SN, Warszawski J, Tinland A. Cumulative incidence of SARS-CoV-2 infection within the homeless population: insights from a city-wide longitudinal study. BMJ Open. 2023 Feb 23;13(2):e065734. doi: 10.1136/bmjopen-2022-065734. PMID 36822808